CLINICAL TRIAL: NCT00807560
Title: Parent-Based Treatment for Pediatric Overweight
Acronym: PO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 07-0216; 1R21HD057394-01 (NIH)
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Adolescents; Family Therapy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FBT-PO (Experimental): Family Based Therapy for Pediatric Overweight.
  Interventions: Behavioral: FBT-PO
- NEC-control (Active Comparator): Nutritional Educational Control Condition (NEC).
  Interventions: Behavioral: NEC

INTERVENTIONS:
Behavioral: FBT-PO — The goal of FBT-PO is to resolve the eating disorder and return the patient to healthy psychosocial and physiological developmental trajectories through active family involvement across three treatment phases.
  Other Names: Family Based Therapy for Pediatric Overweight
  Arms: FBT-PO
Behavioral: NEC — Families assigned to NEC will receive a minimal nutrition and physical activity education curriculum across 16 sessions over 24 weeks.
  Other Names: Nutritional Educational Control Condition
  Arms: NEC-control

SUMMARY:
The purpose of this study is to determine whether a parent/guardian intervention for adolescent overweight/obesity more effective than a nutritional counseling education curriculum for reducing body mass index z-score (BMI Z-score) and related outcomes.

DETAILED DESCRIPTION:
Rates of pediatric overweight (PO) among Americans are increasing and associated with significant psychological, social, quality of life, and health related outcomes. Because of the broad mental and physical health implications of PO and the difficulty in sustaining weight loss as an adult, it is of interest to find successful methods of weight loss and/or prevention of weight gain for obese children and adolescents. The family unit is a logical and empirically supported point of intervention for PO. Interventions on this level have shown good long term efficacy in young children, but there is very little research on adolescent family intervention. Within the eating disorder literature, there is growing support for the efficacy of family-based interventions (FBI) for adolescents. Given its trans-developmental applicability, focus on family as the unit of intervention, and utility in creating a healthy eating environment, FBI is a logical candidate for adaptation to intervention for PO and intervention for at-risk for overweight youth (FBI-PO). The core of the current project is to test the feasibility and efficacy of an adapted FBI manual for adolescent overweight and at-risk for overweight in an outpatient eating and weight disorders clinic and compare this modality to a minimal nutritional educational control (NEC) condition.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13-17
* Male and female
* Living with at least one parent or guardian who is willing to participate in treatment
* A BMI percentile >85% for gender and age (e.g., overweight or at risk for overweight)

Exclusion Criteria:

* Current psychotic illness
* Current alcohol/drug dependence
* Active suicidality
* Eating disorders (e.g., binge eating disorder)
* History of bariatric surgery
* Medication associated with significant weight changes (e.g., antipsychotics)
* Serious medical or physical conditions resulting in significant weight changes (e.g., pregnancy, genetic disorders).
* Complications of obesity that contraindicate moderate physical activity (e.g. orthopedic disorders)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Loeb, PH.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - The University of Chicago, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- FBT-PO: Family Based Therapy for Pediatric Overweight.
  FBT-PO : The goal of FBT-PO is to resolve the eating disorder and return the patient to healthy psychosocial and physiological developmental trajectories through active family involvement across three treatment phases.
- NEC- Control: Nutritional Educational Control Condition (NEC).
  NEC : Families assigned to NEC will receive a minimal nutrition and physical activity education curriculum across 16 sessions over 24 weeks.
Period: Overall Study
Arm/Group | FBT-PO | NEC- Control
Started | 38 | 39
Completed | 38 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NEC-control: Nutritional Educational Control Condition
- Total: Total of all reporting groups
Arm/Group | FBT-PO | NEC-control | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.52) | 15.2 (1.6) | 15.1 (1.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  United States | 38 | 39 | 77

OUTCOME MEASURES:

1. Secondary Outcome: Percent Completion
Description: Percent of participants who completed the trial to assess feasibility and retention in the trial
Time Frame: at 44 weeks
Measure: Number; unit: percentage of participants
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 38 | 39
percentage of participants | 34.2 | 28.2

2. Secondary Outcome: Waist Measurement
Description: Waist measurement in inches. This is not a primary outcome variable.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 38 | 39
inches | 42.0 (3.5) | 44.5 (4.6)

3. Secondary Outcome: Waist Measurement
Description: Waist measurement in inches. This is not a primary outcome variable.
Time Frame: up to 44 weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 8 | 9
inches | 41.7 (3.6) | 45.3 (3.9)

4. Secondary Outcome: Hip Measurement
Description: Hip measurement in inches. This is not a primary outcome variable.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 38 | 39
inches | 47.1 (10.4) | 49.6 (4.8)

5. Secondary Outcome: Hip Measurement
Description: Hip measurement in inches. This is not a primary outcome variable.
Time Frame: up to 44 weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 8 | 9
inches | 47.3 (11.0) | 50.3 (4.5)

6. Secondary Outcome: Height
Description: This variable informs the calculation of the outcome variable of BMI Z score.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 38 | 39
inches | 65.7 (3.0) | 64.7 (2.79)

7. Primary Outcome: BMI Z Score
Description: Z-score was calculated using the Baylor College of Medicine Children's Nutrition Research Center's online BMI calculator (https://www.bcm.edu/research/centers/childrens-nutrition-research-center/bodycomp/bmiz2.html).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 38 | 39
Z-score | 2.3 (.41) | 2.4 (.25)

8. Secondary Outcome: Height
Description: This variable informs the calculation of the outcome variable of BMI Z score.
Time Frame: up to 44 weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 13 | 11
inches | 66.1 (2.7) | 64.8 (2.9)

9. Secondary Outcome: Weight
Description: This variable informs the calculation for the outcome variable of BMI Z score.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 38 | 39
pounds | 213.1 (31.9) | 227.8 (63.8)

10. Secondary Outcome: Weight
Description: This variable informs the calculation of the outcome variable of BMI z score.
Time Frame: up to 44 weeks
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 13 | 11
pounds | 213.3 (33.2) | 233.0 (64.1)

11. Secondary Outcome: BMI
Description: Body Mass Index: this variable informs the calculation of the outcome variable of BMI z-score.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 38 | 39
kg/m^2 | 35.3 (5.5) | 36.6 (6.6)

12. Secondary Outcome: BMI
Description: Body Mass Index: this variable informs the calculation of the primary outcome variable of BMI z-score.
Time Frame: up to 44 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 13 | 11
kg/m^2 | 34.5 (5.2) | 38.7 (9.0)

13. Secondary Outcome: BMI Percentile
Description: Body Mass Index percentile. This is not a primary outcome variable.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 38 | 39
percentile | 98.0 (2.4) | 99.0 (1.1)

14. Primary Outcome: BMI Z Score
Description: as for outcome 7
Time Frame: up to 44 weeks
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 13 | 9
Z-score | 2.2 (0.4) | 2.4 (.12)

15. Secondary Outcome: BMI Percentile
Description: Body Mass Index percentile. This is not a primary outcome variable.
Time Frame: up to 44 weeks
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | FBT-PO | NEC-control
Number analyzed (Participants) | 13 | 9
percentile | 98.3 (2.2) | 99.2 (0.3)

ADVERSE EVENTS:
Arm/Group | FBT-PO | NEC- Control
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 0/38 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes